CLINICAL TRIAL: NCT03737760
Title: Multimodal Imaging of Brain Activity to Investigate Walking and Mobility Decline in Older Adults
Brief Title: "Mind in Motion": Multimodal Imaging of Brain Activity to Investigate Walking and Mobility Decline in Older Adults
Status: Completed | Type: Observational
Sponsor: University of Florida (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Other Study IDs: IRB201802227-N; 1U01AG061389-01 (NIH); OCR19439 (Other: University of Florida); P30AG059297 (NIH); IRB201900001 (Other: UF IRB-01 SubStudy); IRB202201585 (Other: UF IRB-01 SubStudy)
Record Dates: First submitted 2018-11-08; First posted 2018-11-09 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Effect of Age-related Changes in the Brain on Walking Ability
Keywords: walking; aging; brain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Older Adults: Community-dwelling men and women age 70+ years
- Younger Adults: Healthy young adults, age 20-40 years for baseline assessments only

SUMMARY:
The objective of this study is to determine the central neural control of mobility in older adults by acquiring data with multiple modalities of neuroimaging (EEG, fNIRS, MRI) and associating these data with a comprehensive set of diverse mobility outcomes (clinic-based walking, complex walking and community mobility measures).

DETAILED DESCRIPTION:
This study is a longitudinal, prospective cohort study with a follow-up period of 1.2 - 3.5 years, dependent on when the participant enrolls. Participants will be assessed at baseline, and then every six months for 3.5 years or until the study ends, whichever comes first.

The investigators plan to enroll 200 community-dwelling men and women age 70+ years.

ELIGIBILITY:
Inclusion Criteria for Older Adults:

* Community dwelling men and women 65+ years old, or 60+ for individuals who belong to underrepresented racial or ethnic groups;
* Short Physical Performance Battery (SPPB) <10 (45% of the sample will have an SPPB < 8) for moderate to low functioning older adults; SPPB>=10 for high functioning older adults
* Able to complete the 400 m walk test within 15 minutes without sitting or the help of another person and without a walker, a cane is allowed
* Willingness to undergo all testing procedures
* English speaking
* Willingness to be enrolled for 1.25 to 3.5 years, depending on enrollment date.

Inclusion Criteria for Young Adults:

* Healthy men and women aged 20-40 years old
* Willingness to undergo all testing procedures
* English speaking

Exclusion Criteria for all participants:

* Significant medical event requiring hospitalization in the past 6 months that has the potential to contaminate data being collected (fracture, hospitalization etc.);
* Severe visual impairment or corrected visual acuity less than 20/40, which would preclude completion of the assessments;
* Not meeting MRI eligibility (e.g. metal implants, pacemaker, etc.)
* Clinically diagnosed vestibular dysfunction;
* Unwilling or unable to do an over-ground version of the uneven terrain task without assistive device;
* Develops chest pain or severe shortness of breath during physical stress;
* Stroke or other brain injury within the past three years;
* Current presence of motor deficits caused by a stroke or other brain injury;
* Diagnosis of dementia or taking cholinesterase inhibitors (Aricept, Exelon, Razadyne, Namenda, or Namzaric);
* Any major ADL disability (unable to feed, dress, bath, use the toilet, or transfer);
* Report of severe lower extremity pain that significantly limits mobility;
* Diagnosis or treatment for rheumatoid arthritis;
* Lives in a nursing home; persons living in assisted or independent housing will not be excluded;
* Receiving physical therapy for gait, balance, or other lower extremity training;
* Known neuromuscular disorder or overt neurological disease (e.g. Multiple Sclerosis, Rhabdomyolysis, Myasthenia Gravis, Ataxia, Apraxia, post-polio syndrome, mitochondrial myopathy, Parkinson's Disease, ALS etc.)
* Unable to communicate because of severe hearing loss or speech disorder;
* Planned surgical procedure or hospitalization in the next 12 months (e.g., joint replacement, CABG);
* Severe pulmonary disease, requiring the use of supplemental oxygen;
* Terminal illness, as determined by a physician;
* Severe cardiac disease, including NYHA Class III or IV congestive heart failure, clinically significant aortic stenosis, recent history of cardiac arrest, use of a cardiac defibrillator, or uncontrolled angina;
* Is planning to move out of the area in next year or leave the area for >6 mos during follow-up;
* Other significant conditions that would impact safety and/or compliance to the protocol (e.g. renal failure on hemodialysis, psychiatric disorder-bipolar, schizophrenia, excessive alcohol intake etc.);

  -Actively enrolled in an intervention study
* Use of walker or wheel chair;
* Artificial hair covering the scalp such as a wig or toupee
* Failure to provide informed consent;
* Transaminases >twice upper limit of normal;
* Hemoglobin <10 g/dL;
* Investigator discretion based on safety or compliance concerns

  -Temporary exclusion criteria (participant may be eligible if these issues are resolved in the future):
* Abnormalities in blood chemistry parameters as defined above;
* Severe hypertension, e.g., SBP > 200, DBP > 110 mmHg;
* Uncontrolled diabetes or hyperglycemia (fasting blood glucose > 126 mg/dl or hemoglobin A1C > 6.5%)
* Other temporary events that would influence participation (e.g. episodic health event, sick spouse, bereavement, or recent move);
* Other conditions identified with medical history at enrollment that places the participant at risk for participation.

Ages: 20 Years to 110 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Older adults (age 70+) and young adults (age 20-40)
Sampling Method: Non-Probability Sample
Enrollment: 279 (Actual)
Dates: Start 2019-04-19 (Actual); Primary Completion 2025-05-31 (Actual); Study Completion 2025-05-31 (Actual)

PRIMARY OUTCOMES:
Brain activity during walking | Baseline up to 42 months
  Changes in brain activity during complex walking (uneven terrain), assessed longitudinally for up to 3.5 years

CONTACTS AND LOCATIONS:
Overall Officials: David Clark, ScD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States